CLINICAL TRIAL: NCT02280395
Title: A Phase I/II Double-Blind, Randomized, Controlled Study to Evaluate the Safety and Efficacy of RUT058-60 Lavage Following Abdominal Surgery as an Adjunctive Therapy to Prophylactic Systemic Antibiotics
Brief Title: A Phase I/II Double-Blind, Randomized, Controlled Study to Evaluate the Safety and Efficacy of RUT058-60
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Company merger resulted in business decision to terminate the study.
Sponsor: Pulmatrix Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CP02-117838
Record Dates: First submitted 2014-10-26; First posted 2014-10-31 (Estimated); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Postoperative Wound Infection-deep; Post Operative Wound Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Therapeutic Irrigation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RUT058-60 (Experimental)
  Interventions: Drug: RUT058-60
- Sterile Saline for Irrigation (Placebo Comparator)
  Interventions: Drug: Sterile saline for irrigation

INTERVENTIONS:
Drug: RUT058-60 — Prior to closure of the abdomen at the end of the surgical repair, each subject will undergo lavage with approximately 900 mL of RUT058-60 administered as two 400 mL intra-abdominal (peritoneal) lavages and one 100 mL lavage above the fascia.
  Arms: RUT058-60
Drug: Sterile saline for irrigation — Prior to closure of the abdomen, each subject will undergo lavage with approximately 900 mL of sterile saline administered as two 400 mL intra-abdominal (peritoneal) lavages and one 100 mL lavage above the fascia.
  Arms: Sterile Saline for Irrigation

SUMMARY:
This is a double-blind, randomized, parallel-group, controlled, multi-center study to evaluate the safety and efficacy of RUT058-60 (Group A) as an intra-cavity lavage compared to sterile saline (Group B) in adult subjects undergoing abdominal surgery.

DETAILED DESCRIPTION:
Post-surgical site infections account for approximately 20% of total healthcare-associated infections (HAI), making surgical site infections the most common HAI in US hospitals. Despite the routine use of prophylactic systemic antibiotics and improvements in surgical techniques, surgical site infections continue to be associated with significant morbidity, reduction in quality of life and overall cost following abdominal surgery.

Ruthigen is conducting this Phase I/II clinical study to evaluate the safety and potential efficacy of RUT058-60 in preventing surgical deep incisional and organ space infection in subjects undergoing abdominal surgery as an adjunctive therapy to prophylactic systemic antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent to participate in the study and authorization to release health information
* Males or females that are at least 2-years post-menopausal or surgically sterile; 18 to 75 years of age at screening
* Good general health defined as an ASA Physical Status score of moderate or 1 (healthy) or 2 (mild systemic illness), no clinically significant abnormal findings which, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results. Clinical laboratory values ->/+20% outside the normal range may be deemed acceptable
* Willing and able to follow study instructions and available to complete all study requirements and visits
* Scheduled to undergo a planned, non-emergent abdominal surgical procedure involving an open incision of ≥7 cm and ≤35 cm in length. Eligible surgeries include, but may not be limited to: left hemicolectomy, right hemicolectomy, transverse colectomy, total abdominal colectomy with ileorectal anastomosis, lower anterior surgeries, abdominoperineal resection, Ileostomy closures and HARTMAN take down.

Exclusion Criteria:

* Tumor debulking, contaminated surgeries (e.g., extruded bowel) minimally invasive procedures, Caesarian section and hysterectomy
* Laparoscopic appendectomy
* History of allergy or sensitivity to any components of the investigational product
* Body mass index [BMI] >40
* American Society of Anesthesiologists' (ASA) Classification of Physical Status score ≥ 3 (severe systemic illness)
* Evidence preoperatively, of any of the following: sepsis, severe sepsis, or septic shock, or a history of delayed wound healing
* Current surgical site infection (superficial, deep incisional or organ/space) secondary to previous laparotomy/ laparoscopy, or from any other cause
* Receiving any oral or intravenous antibiotics within 1-week prior to Baseline Day 0. Prophylactic antibiotics for dental or other brief procedures are acceptable. Pre-surgical administration of antibiotics is required as part of surgery preparation.
* Preoperative evaluation suggests intra-abdominal process that might preclude full closure of the skin
* History of chemotherapy within 4-weeks or radiation therapy within 4-weeks prior to Baseline
* Terminal illness with life expectancy of less than 6 months from Baseline
* Current smokers, malnourished subjects, subjects with diabetes or uncontrolled serum glucose
* History of major organ transplantation, including bone marrow transplantation
* History of laparotomy within 60-days prior to Baseline
* Preoperative pain threshold (PT) or international normalized ration (INR) >2 x upper limit of normal
* Taking the following concomitant medications within 2 weeks prior to Baseline; systemic steroids or other anti-inflammatory/immunosuppressive medication, or have a history of a current immunosuppressive condition or immune deficiency.Anti-inflammatory medications taken pro re nata (PRN) are allowed per institution/ investigator restriction
* HIV patients or patients with Hepatitis B or C
* Prosthetic cardiac valve or joint prostheses and any potential for remote body site infection
* Medically significant cardiac arrhythmia, or prolonged corrected QT interval (QTc) interval >450 msec
* An ATE (MI, cerebrovascular attack [CVA], TIA), venous thromboembolic event [VTE] (e.g., deep vein thrombosis [DVT], PE), within 12 months of Baseline
* Increased hemorrhage risk (e.g., coagulation disorders)
* Women of child bearing potential (WOCBP) or females that are pregnant, nursing, or planning a pregnancy during the study
* Current enrollment in an investigational drug or device study or participation in such a study within the last 30 days prior to Baseline (Day 0)
* Evidence of active uncontrolled infection or unstable or severe intercurrent medical conditions. All subjects must be afebrile at Baseline (i.e., <38.0° Celsius [C])
* History of stage IV cancer*, other clinically significant renal, hepatic, neurologic, hematologic, respiratory, psychiatric, cardiovascular, infectious disease, psychological condition or social situation which, in the opinion of the Investigator, puts the subject at significant risk, could confound the study results, or may interfere significantly with the subject's participation in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability will be determined by nature and incidence of adverse events and clinical laboratory values compared to saline control group. Wound site physical inspection tabulated result compared to saline control group. | 28 Days

SECONDARY OUTCOMES:
Potential efficacy will be determined by the proportion of subjects who do not develop a surgical deep incisional or organ/space infection by Day 28 post-application compared to the saline control group. | 28 Days
  In each of the two groups, the proportion of subjects who are deep incisional and organ/space infection-free will be estimated, along with a two-sided, 90% exact binomial confidence interval for the true rate in each group.

OTHER OUTCOMES:
Exploratory Analysis- Overall length of hospital stay | 28 Days
Exploratory Analysis- Readmission to the hospital within the first 28-days post-operative procedure | 28 Days
Exploratory Analysis- Incisional wound healing time frame | 28 Days

CONTACTS AND LOCATIONS:
Overall Officials: Traci Hedrick, MD, Principal Investigator — University of Virginia; Timothy I Melson, MD, Principal Investigator — Shoals Medical Trials, Helen Kellar Hospital; Harold Minkowitz, MD, Principal Investigator — BJJS Corporation, Memorial Hermann Memorial Medical Center; Paul Rider, MD, Principal Investigator — University of South Alabama Medical Center; Sonia Ramamoorthy, MD, Principal Investigator — University of California, San Diego; AnaMaria Garza, MD, Principal Investigator — PVMDI, Glendale Memorial (Dignity Health)
Locations (4):
- United States (4):
  - University of South Alabama Medical Center, Mobile, Alabama
  - University of California, San Diego, Thornton Hospital, La Jolla, California
  - BJJS, Corp., Memorial Hermann Memorial Medical Center, Houston, Texas
  - University of Virginia, Charlottesville, Virginia